CLINICAL TRIAL: NCT01461824
Title: Relationship Between Drug Exposure and DNA Markers With Depot Medroxyprogesterone Acetate-associated Side Effects in Adolescents
Brief Title: Drug Exposure and Depot Medroxyprogesterone Acetate (DMPA) in Adolescent Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Andrea Bonny, Assistant Professor, Department of Pediatrics, The Ohio State University, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB11-00583
Record Dates: First submitted 2011-10-21; First posted 2011-10-28 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Weight Gain; Disorder of Bone Density and Structure, Unspecified; Uterine Bleeding
Keywords: Birth Control; Contraceptive Methods; Female Contraception; Weight Gain; Bone Density
MeSH Terms: conditions — Weight Gain; Uterine Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 150 mg DMPA (Active Comparator): Depot medroxyprogesterone acetate (DMPA) 150 mg every 12 weeks IM
  Interventions: Drug: Depot medroxyprogesterone acetate (DMPA)
- 104mg DMPA (Experimental): Depot medroxyprogesterone acetate (DMPA) 104 mg every 12 weeks IM
  Interventions: Drug: Depot medroxyprogesterone acetate (DMPA)
- 75mg DMPA (Experimental): Depot medroxyprogesterone acetate (DMPA) 75 mg every 12 weeks IM
  Interventions: Drug: Depot medroxyprogesterone acetate (DMPA)

INTERVENTIONS:
Drug: Depot medroxyprogesterone acetate (DMPA) — 75mg, 104mg and 150mg DMPA, IM, every 12 weeks for 12 months
  Other Names: Generic Depo Provera manufactured by Greenstone, LLC

SUMMARY:
The investigators are doing this study to look at how different doses of the Depot medroxyprogesterone acetate (DMPA) shot effect weight gain and bone mineral density in teens. The investigators hope that what the investigators learn from this study will be used to develop ways to keep girls from gaining weight or losing bone density when receiving DMPA.

DETAILED DESCRIPTION:
Depot medroxyprogesterone acetate (DMPA) is a generic form of the DepoProvera® shot. When receiving the birth control shot some girls gain a lot of weight while others do not. Some girls also lose bone mineral density (BMD). Bone mineral density is the amount of weight and thickness of the bones.

In this study 1 of 3 doses of DMPA will be given as an injection into the muscle in the arm. The 150mg dose is approved for use in this age group by the Food and Drug Administration (FDA) when given into the muscle. The 104mg dose is approved for use in this age group by the FDA only when given under the skin therefore it is considered experimental. The 75mg dose is also considered experimental as this dose is not FDA approved regardless of how it is given.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-21 years
2. Healthy, post-menarcheal female
3. Self-selected to initiate depot medroxyprogesterone acetate (DMPA)
4. Willingness to use a barrier method of contraception in addition to DMPA

Exclusion Criteria:

1. Chronic disease known to affect weight or bone mineral density (BMD) (e.g. diabetes, kidney)
2. Use of medication known to affect weight or BMD (e.g. corticosteroids)
3. DMPA use within the past 12 months
4. Pregnancy within the past 6 months
5. Etonogestrel implant, levonorgestrel-releasing intrauterine system or combined estrogen/progesterone contraceptive use within the past 30 days (OC, patch, vaginal ring)
6. Weight exceeding 450 lbs
7. Need for confidential contraceptive care for individuals < 18 years of age.

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2011-09; Primary Completion 2015-04 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bonny, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 150 mg DMPA | 104mg DMPA | 75mg DMPA
Started | 12 | 11 | 11
Completed | 10 | 7 | 8
Not Completed | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 150 mg DMPA | 104mg DMPA | 75mg DMPA | Total
Number analyzed (Participants) | 12 | 11 | 11 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.6 (2.1) | 18.3 (2.65) | 19.0 (2.43) | 18.6 (2.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 11 | 34
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 2 | 4 | 13
  White | 5 | 9 | 7 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Lumbar Spine Bone Mineral Density (BMD) From Baseline to 48 Weeks
Description: Lumbar spine bone mineral density measured at baseline and 48 weeks. Percent change over this time was calculated.
Time Frame: Percent change from baseline to 48 Weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 150 mg DMPA | 104mg DMPA | 75mg DMPA
Number analyzed (Participants) | 8 | 7 | 10
percent change | -4.0 (2.76) | -3.1 (1.84) | -0.6 (5.91)

2. Primary Outcome: Proportion of Participants With >5% Weight Gain at 24 Weeks
Description: Individual subjects will be assessed after their Week 24 visit.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg DMPA | 104mg DMPA | 75mg DMPA
Number analyzed (Participants) | 8 | 9 | 10
Participants | 1 | 2 | 2

3. Secondary Outcome: Percent Change in Total Hip BMD From Baseline to 48 Weeks
Description: Total hip bone mineral density was assessed at baseline and 48 weeks. Percent change from baseline to 48 weeks was calculated.
Time Frame: Percent change from baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 150 mg DMPA | 104mg DMPA | 75mg DMPA
Number analyzed (Participants) | 8 | 7 | 10
Percent change | -3.0 (3.22) | -1.6 (2.53) | -0.1 (5.07)

ADVERSE EVENTS:
Time Frame: Up to 48 weeks
Description: Solicited at each visit
Groups:
- 150 mg DMPA: Depot medroxyprogesterone acetate (DMPA):150mg DMPA, IM, every 12 weeks for 12 months
- 104 mg DMPA: Depot medroxyprogesterone acetate (DMPA):104mg DMPA, IM, every 12 weeks for 12 months
- 75 mg DMPA: Depot medroxyprogesterone acetate (DMPA):75mg DMPA, IM, every 12 weeks for 12 months
Arm/Group | 150 mg DMPA | 104 mg DMPA | 75 mg DMPA
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 8/12 | 11/11 | 10/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 150 mg DMPA (N=12) | 104 mg DMPA (N=11) | 75 mg DMPA (N=11)
Headache (Nervous system disorders) | 3 | 3 | 3
Upper respiratory infection (Infections and infestations) | 4 | 8 | 7
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Lip infection (Infections and infestations) | 0 | 1 | 1 — Cold sore
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Viral infection not specified (Infections and infestations) | 2 | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0 | 1 — Contact dermatitis
Uterine pain (Reproductive system and breast disorders) | 2 | 1 | 4 — Cramping
Urinary tract infection (Reproductive system and breast disorders) | 0 | 1 | 2
Irregular menstruation (Reproductive system and breast disorders) | 2 | 3 | 2
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vaginal pain (Reproductive system and breast disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vaginal infection (Reproductive system and breast disorders) | 0 | 0 | 1
Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Bloating (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No